CLINICAL TRIAL: NCT04657172
Title: A Phase 3 Study of the Safety and Efficacy of 1% and 2% Pilocarpine Ophthalmic Solutions Administered With the Optejet® Microdose Dispenser for Temporary Improvement of Near Vision in Adults With Presbyopia
Brief Title: Safety & Efficacy of Pilocarpine Eye Solutions for Temporary Improvement of Near Vision in Presbyopic Adults
Acronym: VISION-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eyenovia Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EYN-PRS-PI-31
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pilocarpine 1% Solution (Experimental): 1% pilocarpine ophthalmic solution administered with the Optejet dispenser
  Interventions: Drug: Pilocarpine Ophthalmic
- Pilocarpine 2% Solution (Experimental): 2% pilocarpine ophthalmic solution administered with the Optejet dispenser
  Interventions: Drug: Pilocarpine Ophthalmic
- Placebo Solution (Placebo Comparator): Placebo ophthalmic solution administered with the Optejet dispenser
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pilocarpine Ophthalmic — Pilocarpine 1% or 2% ophthalmic solution administered with the Optejet microdose dispenser
  Other Names: MicroLine
  Arms: Pilocarpine 1% Solution; Pilocarpine 2% Solution
Drug: Placebo — Vehicle ophthalmic solution administered with the Optejet microdose dispenser
  Arms: Placebo Solution

SUMMARY:
Volunteer participants are evaluated for eligibility during a Screening Visit; those meeting study inclusion/exclusion criteria are scheduled for 3 treatment visits. At each treatment visit, 1 of the 3 study solutions is self-administered to both eyes. Afterwards, efficacy and safety assessments are performed over a 3-hour period.

ELIGIBILITY:
Primary Inclusion Criteria:

* Poor near vision impacting daily living that requires near correction
* Best-corrected distance visual acuity (BCDVA) of 0.0 logMar or better
* Manifest refraction spherical equivalent ≥ -2.00 Diopters (D) and ≤ +2.00 D
* Monocular DCNVA between 0.4 and 0.7 logMAR, inclusive

Primary Exclusion Criteria:

* Diagnosis of glaucoma or ocular hypertension
* Narrow iridocorneal angles
* History of intraocular surgery, refractive surgery, laser treatment, or iris surgery
* Clinically significant abnormality of cornea, lens, retina, ciliary body, or iris
* Presence/history of a severe/serious ocular condition or any other unstable medical condition
* Presence or history of manifest strabismus, amblyopia, or nystagmus
* Current active eye disease for which topical or systemic ophthalmic medication is necessary, except for dry eye syndrome managed using artificial tears
* Clinically significant external ocular inflammation within 30 days of Screening Visit
* Current use or history of rigid gas permeable (RGP) contact lens use within 30 days of Screening Visit
* Known pilocarpine allergy or contraindication to use of pilocarpine
* Presence or history of congenital heart anomaly, valve disease, or other cardiac disease
* Disabling arthritis or limited motor coordination that would limit the subject's ability to self-administer study solution using the Optejet

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects gaining ≥ 15 letters in mesopic, high contrast, binocular distance corrected near visual acuity (DCNVA) | 120 minutes post-dosing
  The proportion of subjects gaining ≥ 15 letters in mesopic, high contrast, binocular DCNVA as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Tsontcho (Sean) Ianchulev, MD, MPH, Study Chair — Eyenovia Inc.
Locations (9):
- United States (9):
  - VISION-1 Study Site #21, Azusa, California
  - VISION-1 Study Site #52, Newport Beach, California
  - VISION-1 Study Site #54, Fort Collins, Colorado
  - VISION-1 Study Site #53, Orlando, Florida
  - VISION-1 Study Site #50, New York, New York
  - VISION-1 Study Site #17, High Point, North Carolina
  - VISION-1 Study Site #22, Raleigh, North Carolina
  - VISION-1 Study Site #51, Cranberry Township, Pennsylvania
  - VISION-1 Study Site #03, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No